CLINICAL TRIAL: NCT00706576
Title: Treatment of Unresectable Hepatocellular Cancer With Opioid Growth Factor: a Phase I Study
Brief Title: Treatment of Unresectable Hepatocellular Cancer With Opioid Growth Factor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Eric Kimchi, Associate Professor of Surgical Oncology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26336
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Hepatocellular Cancer
Keywords: Hepatocellular cancer; HCC; Opioid growth factor; OGF; Cirrhosis
MeSH Terms: conditions — Liver Neoplasms; Fibrosis | interventions — Enkephalin, Methionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infusion of opioid growth factor (Experimental): Volunteers will be treated with an intravenous infusion of opioid growth factor(OGF) starting at 100 µg/kg with a 50 µg/kg dose escalation with each succeeding group. The investigational drug, OGF, will be diluted in sterile saline to its appropriate concentration based upon the body weight of the volunteer and administered in a volume of 60 ml over 45 minutes (rate of 2 ml/min)
  Interventions: Drug: Infusion of opioid growth factor

INTERVENTIONS:
Drug: Infusion of opioid growth factor — Volunteers will be treated with an intravenous infusion of opioid growth factor(OGF) starting at 100 µg/kg with a 50 µg/kg dose escalation with each succeeding group. The investigational drug, OGF, will be diluted in sterile saline to its appropriate concentration based upon the body weight of the volunteer and administered in a volume of 60 ml over 45 minutes (rate of 2 ml/min)
  Other Names: OGF; [Met5]-enkephalin

SUMMARY:
Hepatocellular cancer, one of the world's most deadly tumors, is associated with chronic liver injury and cirrhosis. With the increasing occurrence of viral hepatitis, the incidence of this cancer in the United States continues to rise. Surgical resection offers the only hope for cure; but sadly, few patients are candidates for surgery due to their liver disease. Liver transplant can be an effective treatment, but due to a scarcity of organs, most patients do not qualify for this therapy either. Patients who are not candidates for these procedures have very few therapeutic options as chemotherapy and radiation have little efficacy. New therapies are desperately needed.

Opioid Growth Factor (OGF) inhibits the growth of a number of cancer lines in vitro by a receptor-mediated mechanism. In pancreatic cancer this phenomenon has been well defined not only in vitro but in animal models. Based upon these findings, a phase I trial has been conducted demonstrating that OGF can be administered safely to patients with pancreatic cancer. The investigators hypothesize that administration of OGF will inhibit the course of cancer progression in human subjects with unresectable hepatocellular cancer and cirrhosis. As a first step in testing this hypothesis, the investigators propose a phase I trial to study the toxicity and pharmacokinetics of this therapy in patients suffering from inoperable hepatocellular cancer and cirrhosis.

DETAILED DESCRIPTION:
STUDY OBJECTIVES Hepatocellular cancer (HCC) is one of the most prevalent cancers in the world. About 19,160 new cases are anticipated to occur in the US in 2007. Any form of chronic liver injury and cirrhosis predisposes to the development of this malignancy. Worldwide, the most common risk factor is viral hepatitis; in the United States other sources of chronic liver injury such as cirrhosis related to alcohol use are important, but the incidence of viral hepatitis continues to increase. Regardless of the etiology, the only known cure for HCC is surgical resection. Unfortunately, due to associated liver disease and stage of tumor progression at the time of diagnosis, very few patients are candidates for surgical therapy. Chemotherapy has shown very little efficacy in this disease, and radiation is of little value due to associated liver toxicity. New therapies are desperately needed.

Research examining the mechanisms involved in the growth of human cancer has shown that the peptide [Met5]-enkephalin, Opioid Growth Factor (OGF), inhibits growth of a number of cancer lines in vitro. In pancreatic cancer this phenomenon has been well defined not only in vitro but in vivo after transfer of human tumors into nude mice. The suppressive effect on growth by this peptide is by a receptor-mediated mechanism. Based upon these findings, a phase I trial has been conducted studying the effects of OGF in patients with pancreatic cancer. We hypothesize that administration of OGF will inhibit the course of carcinogenic events in human subjects with unresectable hepatocellular cancer and cirrhosis. In order to test this hypothesis we propose a phase I trial to study the toxicity of this therapy in patients suffering from liver disease and cirrhosis addressing the following specific aims:

Specific Aim 1: Determine the maximum-tolerated dose (MTD) of OGF after an intravenous infusion in patients suffering from HCC. While the MTD has been determined for patients suffering from pancreatic cancer, it is unclear that these results will hold true in patients with HCC who suffer from liver insufficiency and cirrhosis. For this reason we will conduct a dose-finding trial that contains dose-escalation of OGF. Dose-limiting toxicities will be determined by monitoring liver function, pupillary size & response, respiration, vital signs (orthostatic blood pressure and pulse), gastrointestinal distress, cutaneous flushing, and effects on blood count, glucose and electrolytes.

Specific Aim 2: Study the pharmacokinetics and metabolism of OGF in patients with HCC and cirrhosis by monitoring plasma OGF levels. Blood samples will be collected prior to and at designated intervals after an infusion of the MTD of OGF in cancer patients. OGF plasma levels will be analyzed by performing radioimmunoassay.

The long-term objectives of our research team are to understand the effects of peptide growth factors in patients with HCC and cirrhosis. This phase I trial will be useful in determining the appropriate dose and expected toxicities of OGF in these patients. Our study employs the use of a naturally occurring opioid peptide, which has been shown to inhibit growth of pancreatic cancer in preclinical studies, and to be safely administered to patients with pancreatic cancer.

BACKGROUND AND SIGNIFICANCE Hepatocellular carcinoma (HCC) is the fifth most common malignancy in the world; five hundred thousand people succumb to this malignancy annually. The incidence and mortality rates are almost equal, which demonstrates that very few patients are cured. Any form of chronic liver injury and cirrhosis predisposes to the development of this malignancy. The major risk factors for HCC are chronic hepatitis B virus infection, chronic hepatitis C virus (HCV) infection, and alcoholic cirrhosis.

The only known cure for HCC is surgical resection. The patient's degree of cirrhosis and the anatomic location of tumor determine if partial hepatectomy can be performed. Even at high volume centers specializing in the procedure, operative mortality has been shown to increase from 1% to 14% in the presence of cirrhosis (1). For this reason, resection is usually reserved for patients with Child's A liver function. Multiple lesions do not preclude resection. Intraductal tumors causing obstructive jaundice can be successfully resected. In this situation, it is important to distinguish obstruction from underlying liver disease as the cause of the patient's jaundice.

Total hepatectomy followed by orthotropic liver transplantation is a sensible strategy to treat patients with cirrhosis and cancer, and experience is growing with this approach. As expected, the best results have been recorded in patients who had small HCC discovered incidentally at transplantation performed for liver failure. Lesions smaller than 5 cm treated by transplantation have a significantly better prognosis, and, because organs are scarce, transplantation for HCC us usually limited to this setting. Mazzaferro et al have reported liver transplantation as an effective treatment for small, unresectable HCC in patients with cirrhosis, with 4-year recurrence-free survival of 83%.

Unfortunately, 90% of patients are not suitable for resection or transplantation with a curative intent (2-6), and these patients have very few therapeutic options of proven efficacy. In this setting the prognosis is extremely poor, with median survivals as low as 3 months in high-incidence areas (5-8). No systemic chemotherapeutic regimens have demonstrated significant efficacy. Response rates to single-agent and multidrug protocols, with or without biologic response modifiers, are no better than 20% to 30% (9-12)and randomized trials do not demonstrate a clear survival benefit (13, 14). Recently, sorafenib was shown to increase overall survival, from 7.9 months to 10.7 months, in Child's A patients with hepatocellular cancer (15). External radiation therapy for HCC is ineffective even for palliation (9, 16, 17)because the dose of radiation that can be delivered to the tumor is limited by radiation hepatitis (18, 19). Hepatic intraarterial infusion of cytotoxic agents, aimed at increasing the local concentration of drugs and reducing systemic toxicity (20), and intraarterial embolization, which causes ischemic necrosis of the tumor (21), have been used as palliative treatment either alone or in combination. Chemoembolization is most often employed on the basis of reports of decrease in tumor size in nonrandomized trials (22-26); however, the results of a multi-center randomized trial showed no improvement in overall survival, and significant morbidity with this therapeutic approach (27). Clearly new therapeutic strategies are needed to treat this deadly disease.

Endogenous opioid systems participate in the growth of developing cells and tissues, micro-organisms, tissues that undergo cellular renewal, and in neoplastic cells and tissues (28, 29). A thorough examination of the effects of opioid peptides in pancreatic cancer cells growing in tissue culture revealed that [Met5]- enkephalin, a pentapeptide was the most potent peptide influencing DNA synthesis and growth; in view of its growth factor action, [Met5]-enkephalin has been termed opioid growth factor (OGF). OGF interacts with the OGFr receptor zeta (OGFr) to influence growth. Unlike other opioid receptors, the function (e.g., growth), distribution (neural and non-neural), transient appearance during ontogeny, ligand specificity (i.e., [Met5]- enkephalin), competitive inhibition profile, subcellular location (i.e., nucleus), and the fact that ligands for other known opioid receptors do not influence growth have provided a unique set of characteristics that distinguish the OGFr from other opioid receptors. It has been demonstrated that opioids function as inhibitory growth factors in human pancreatic cancer, both in vitro and in vivo (28, 30).

[Met5]-enkephalin has been safely used in several pilot studies to treat human subjects with cancer. Wybran and Schandene (31) administered [Met5]-enkephalin intravenously to seven previously untreated patients with lung cancer and found significant increases in T-cell immunity (i.e., OK1 0 cells. Leu11 cells, and natural killer cells). Plotnikoff and colleagues (32) administered [Met5]-enkephalin over a period of several months by intravenous infusions at doses of 10 to 60 pg/kg body weight three times weekly to human subjects with advanced melanoma. Plotnikoff and coworkers (33) and Wybran and coworkers (31) have reported improvement in the size and coloration of Kaposi's sarcoma nodules in AIDS patients. In addition, [Met5]-enkephalin increased the number of cytotoxic T-cells and NK cells involved in tumor surveillance. The tumor response in these human studies has been attributed to [Met5]-enkephalin's action on the immune system (31, 34). Most recently, a phase I study has demonstrated that OGF can be delivered safely to patients suffering from advanced pancreatic cancer (30) and is now being given in a phase II trial.

Our research team has demonstrated both the presence and the function of the Opioid Growth Factor (OGF)-OGF receptor (OGFr) system in human hepatocellular carcinoma. First, immunohistochemistry staining of human hepatocellular cell lines SK-Hep-1 and HepG2 cells revealed specific distribution of both OGF and OGFr. Second, OGFr was detected in receptor binding studies, and found to have specific and saturable binding of a single binding site, with binding capacity (Bmax) values of 12.1 +/- 2.7 fmol/mg protein and 9.4 +/- 1.9 fmol/mg protein and binding affinity (Kd) values of 6.1 +/- 1.1 nM and 5.8 +/- 1.5 nM for SK-Hep-1 and HepG2, respectively. Third, in functional assays that monitored the effects of OGF on cell number of human hepatocellular carcinoma cells, a statistically significant suppression in cell growth was found in vitro when SK-Hep-1 cell were cultured in the presence of OGF (appendix 10.7). Based on the previous in vitro and in vivo evidence in pancreatic cancer, as well as with colon cancer, neuroblastoma, and squamous cell carcinoma of the head and neck, as well as the successful Phase I trial of OGF in pancreatic cancer patients, these preliminary data with hepatocellular carcinoma cells are consistent and provide the rationale to test OGF therapy in patients with hepatocellular carcinoma and cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* In this acute dose-finding section of the study, we will enroll patients with HCC and cirrhosis.
* Both male and female patients 18 years of age or older will be eligible.
* Patients with cancer must have a Karnofsky performance rating of at least 50%.
* Patients must have HCC and cirrhosis that is not amenable to current therapies including liver resection, tumor ablation, or liver transplant.
* Patients must be mentally alert and able to give informed consent.
* Female patients who are menopausal, or of childbearing age who are surgically sterile or practicing birth control (chemical or mechanical) are eligible.
* All females of childbearing potential must have a serum pregnancy test upon entry into the study and must take precautions to not become pregnant during the study (from the time of enrollment until 1 week after the infusion of OGF). No corticosteroid or narcotic therapy 24 hrs prior to infusion.
* Volunteers must refrain from alcoholic beverages for 24 hours before, and 24 hours after, the day of infusion.
* If patients have received sorafenib, at least 4 weeks must pass from the last dose.
* At least four weeks must pass from significant surgery and the subject must be physically recovered.

Exclusion Criteria:

* Patients with asthma, chronic obstructive pulmonary disease, unstable cardiovascular diseases (congestive heart failure, symptoms of coronary artery disease, cardiac arrhythmias, poorly controlled hypertension, have suffered a myocardial infarction in the preceding year or have an abnormal EKG) will not be allowed.
* Patients with poorly controlled diabetes, seizure disorders, primary central nervous system (CNS) tumors or known brain metastases are excluded.
* A clinical judgment will be made based on the other criteria and performance status as to the patient's ability to tolerate therapy.
* Serum total bilirubin and international normalized ratio (INR) will be used as markers of liver function in the exclusion criteria as defined in Table 1 (see below).
* Pregnant or nursing women are not eligible.
* Patients requiring antibiotics in the preceding week for a serious infection are not eligible.
* Volunteers may have on the morning of the study one 8 ounce glass of water or juice and toast.
* EKG and laboratory tests will be reviewed to evaluate whether any exclusion criteria are met.
* Those who are not eligible will be notified.

Table 1: Exclusion Criteria

* Leukocyte Count < 3500/μl
* Hemoglobin < 8500/μl
* Blood urea nitrogen (BUN) > 30mg/dl (hydrated)
* Creatinine > 2 mg/dl
* Platlet Count < 55,000/mm3
* INR (unless on coumadin) > 2
* Total Bilirubin > 3.5mg/dl
* Sodium < 130 mmol/L
* Potassium <3.2 mmol/L
* Glucose > 300 or < 60 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with opioid growth factor toxicity | Over the period of infusion and 1 hour after infusion
  primary outcome variable is toxicity and or tolerance to opioid growth factor in patients with hepatocellular cancer

SECONDARY OUTCOMES:
Change in plasma opioid growth factor levels | During the infusion and 1 hour after infusion
  Study the biological kinetics and metabolism of opioid growth factor (OGF) by monitoring plasma OGF levels

CONTACTS AND LOCATIONS:
Overall Officials: Eric T Kimchi, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided